CLINICAL TRIAL: NCT04213846
Title: Personalized Mobile Phone App Intervention: Challenging Alcohol Expectancies to Reduce High-risk Alcohol Use and Consequences
Brief Title: Alcohol & Mobile Phone Study to Reduce High-risk Alcohol Use and Consequences
Acronym: AMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christine Lee, Research Professor, School of Medicine: Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002769; 2R01AA016979-05A1 (NIH)
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Alcohol; Use, Problem
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two conditions (mobile Alcohol Expectancy Intervention and assessment-only control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Alcohol Expectancy Intervention (Experimental): Participants randomized to the intervention condition will receive twice daily intervention messages for three weeks and have access to other psycho-educational alcohol information.
  Interventions: Behavioral: Experimental: Mobile Alcohol Expectancy Intervention
- Assessment-only Control (No Intervention): Participants randomized to the control group will not receive any intervention. They will be an assessment-only control group.

INTERVENTIONS:
Behavioral: Experimental: Mobile Alcohol Expectancy Intervention — Participants randomized to the intervention condition will receive daily intervention messages two times a day for three weeks in the mobile app. The intervention uses participants' own daily responses to personalize messages, when appropriate, that challenges their personal expectations of alcohol's positive effects on mood, social facilitation, and tension reduction, as well as aggression and risk-taking. The intervention messages also focus on intentions to drink and pharmacologically-delayed negative effects. Intervention Messages in general will include feedback based on selected assessment items, weekly summaries generated from the daily assessments, general psycho-educational messages and videos about alcohol, and a toolbox with supplemental information (e.g., personal BAC calculators, resources).
  Arms: Mobile Alcohol Expectancy Intervention

SUMMARY:
The proposed study will develop a smartphone/mobile app intervention that incorporates ecological momentary assessment (i.e., two brief surveys per day) and daily intervention messaging (2 messages per day) for three weeks to target high-risk alcohol use among young adult college students. The intervention mainly focuses on alcohol expectancies, alcohol use, and consequences and the daily associations between these and includes personalized intervention messages based on participants' own event-level expectations and experiences. Other psycho-educational alcohol-related content is also provided over the course of three week intervention. This mobile app intervention will be used in a randomized controlled trial (RCT) comparing young adult college students who receive the intervention with those who only receive assessments via the mobile app.

DETAILED DESCRIPTION:
The purpose of this study is to develop and test a smartphone app that can both collect daily data and deliver a personalized intervention using participants' own event-level, real-world experiences to challenge proximal alcohol expectancies and alter the associations between alcohol expectancies and drinking and consequences. The mobile app intervention will be used in a randomized controlled trial comparing young adult college students who receive the intervention with those who only receive assessments via the mobile app. Assessments include an eligibility survey, baseline assessment, and follow-up assessments occurring 1-, 6-, and 12-months post-intervention.

The goal of the intervention is to target college students' alcohol expectancies (what they believe or expect alcohol's effects to be) and the associations between alcohol expectancies and alcohol use and related consequences. Intervention content will utilize twice daily messages, one in the morning (AM Messages) and one in the late afternoon or early evening (PM Messages). Most PM Messages draw on information collected in the daily assessments (Personalized Messages). Intervention Messages in general will include feedback based on selected assessment items, weekly summaries generated from the daily assessments, general psycho-educational messages and videos about alcohol, and a toolbox with content that supplements information provided in the daily intervention messages.

ELIGIBILITY:
Inclusion Criteria:

* Typically drinking 2+ days/week, having at least 1 occasion of heavy episodic drinking (4+ women/5+ men) in last 2 weeks, having 4 or more negative consequences in the last month, owning a smartphone with a data package, agreeing to install the app on their phone and receive notifications.
* Student at a 2- or 4- year college where recruitment is located

Exclusion Criteria:

* None

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 408 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Lee, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Datasets with cross-sectional and/or longitudinal datasets will be available in Microsoft Excel, where it can be transferred easily to a statistical program such as SAS, Stata, SPSS, or R. Codebooks to assist with data analyses and interpretation will be created and can be shared. We plan to make the datasets available for sharing at the time that the main project findings are published or shortly thereafter. We will share data that do not compromise individuals' rights and privacy available in accordance with the University of Washington (UW) IRB policies. To facilitate replication in other studies, all measures we use are available in the public domain and are popular measures of alcohol use, alcohol-related consequences or alcohol expectancies. For any measure we modify or create for our purposes, we will described in detail (with added items listed) these changes in our published work.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The raw datafile and codebook, which will initially be used for internal study team purposes, will be available for public use after our main aims paper are published; approximately one year of the final year of funding.
  Analytic code will be made available upon request after publication of manuscript.
Access Criteria: Individual researchers can contact the PI for data requests. Researchers can request datasets to replicate published papers and/or for new unpublished analyses unrelated to main study aims. After contacting the PI, researchers will be requested to fill out a questionnaire with respect to data requested and appropriate forms for data sharing. Requests will be reviewed by the PI and co-investigators to determine if analyses are currently underway for the same variables. If not, study documentation and de-identified data will be made available to the requestor.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Assessment-only Control | Mobile Alcohol Expectancy Intervention
Started | 203 | 205
Completed | 181 | 178
Not Completed | 22 | 27
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Lost to Follow-up | 15 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Assessment-only Control | Mobile Alcohol Expectancy Intervention | Total
Number analyzed (Participants) | 203 | 205 | 408
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 203 | 205 | 408
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.78 (1.59) | 20.90 (1.66) | 20.84 (1.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 131 | 260
  Male | 74 | 74 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 30 | 63
  Not Hispanic or Latino | 167 | 169 | 336
  Unknown or Not Reported | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 37 | 39 | 76
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 10 | 3 | 13
  White | 125 | 131 | 256
  More than one race | 16 | 24 | 40
  Unknown or Not Reported | 12 | 6 | 18
Region of Enrollment [Number; unit: participants]
  United States | 203 | 205 | 408
School Type [Count of Participants; unit: Participants]
  4-year college | 153 | 153 | 306
  2-year college | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Daily Drinking Questionnaire - Typical Number of Drinks Per Week
Description: The count of self-reported typical number of drinks consumed per week during the past month
Time Frame: Baseline, 1-month follow-up, 6-month follow-up, and 12-month follow-up
Population: Difference in number analyzed by condition are due to differences in follow-up participation rates and/or items skipped by participants.
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | Assessment-only Control | Mobile Alcohol Expectancy Intervention
Number analyzed (Participants) | 203 | 205
drinks
  Baseline: number analyzed (Participants) | 203 | 204
  Baseline | 13.51 (10.17) | 12.23 (8.49)
  1-month follow-up: number analyzed (Participants) | 188 | 192
  1-month follow-up | 10.70 (10.29) | 8.95 (7.76)
  6-month follow-up: number analyzed (Participants) | 183 | 169
  6-month follow-up | 9.46 (9.47) | 9.06 (8.46)
  12-month follow-up: number analyzed (Participants) | 178 | 172
  12-month follow-up | 9.91 (11.22) | 8.81 (7.83)
Statistical Analysis 1: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 1-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — Generalized linear mixed model was estimated using a sample of N=408 with a Condition × 1-Month Follow-Up interaction. Assessment-only control was the reference category for Condition, and Baseline was the reference category for 1-Month Follow-Up; p = 0.34, Generalized linear mixed model; Models controlled for sex, age, and college type (2-year vs. 4-year) and used a Poisson error distribution; Count/Rate Ratio = 0.94, 95% CI 2-sided [0.81 to 1.07]
Statistical Analysis 2: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 6-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — Generalized linear mixed model was estimated using a sample of N=408 with a Condition × 6-Month Follow-Up interaction. Assessment-only control was the reference category for Condition, and Baseline was the reference category for 6-Month Follow-Up; p = 0.37, Generalized linear mixed model; Models controlled for sex, age, and college type (2-year vs. 4-year) and used a Poisson error distribution; Count/Rate Ratio = 1.09, 95% CI 2-sided [0.91 to 1.30]
Statistical Analysis 3: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 12-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — Generalized linear mixed model was estimated using a sample of N=408 with a Condition × 12-Month Follow-Up interaction. Assessment-only control was the reference category for Condition, and Baseline was the reference category for 12-Month Follow-Up; p = 0.80, Generalized linear mixed model; Models controlled for sex, age, and college type (2-year vs. 4-year) and used a Poisson error distribution; Count/Rate Ratio = 1.02, 95% CI 2-sided [0.85 to 1.23]

2. Primary Outcome: Peak Estimated Blood Alcohol Concentration (Peak eBAC)
Description: The eBAC reached during the heaviest drinking episode during the past month based on self-reported number of drinks, sex, and hours drinking
Time Frame: Baseline, 1-month follow-up, 6-month follow-up, and 12-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | Assessment-only Control | Mobile Alcohol Expectancy Intervention
Number analyzed (Participants) | 203 | 205
grams per deciliter
  Baseline: number analyzed (Participants) | 201 | 203
  Baseline | 0.19 (0.14) | 0.16 (0.10)
  1-month follow-up: number analyzed (Participants) | 187 | 190
  1-month follow-up | 0.15 (0.11) | 0.14 (0.11)
  6-month follow-up: number analyzed (Participants) | 183 | 168
  6-month follow-up | 0.14 (0.12) | 0.13 (0.10)
  12-month follow-up: number analyzed (Participants) | 178 | 170
  12-month follow-up | 0.14 (0.11) | 0.13 (0.10)
Statistical Analysis 1: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 1-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.75, Generalized linear mixed model; Models controlled for sex, age, college type and used a Poisson error distribution. Peak eBAC multiplied by 100 and rounded up to the nearest integer; Count/Rate Ratio = 1.02, 95% CI 2-sided [0.88 to 1.20]
Statistical Analysis 2: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 6-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.72, Generalized linear mixed model; [statistical method as in outcome 2, analysis 1]; Count/Rate Ratio = 1.04, 95% CI 2-sided [0.86 to 1.25]
Statistical Analysis 3: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 12-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 3]; p = 0.91, Generalized linear mixed model; [statistical method as in outcome 2, analysis 1]; Count/Rate Ratio = 1.01, 95% CI 2-sided [0.85 to 1.21]

3. Primary Outcome: Number of Heavy Episodic Drinking Days
Description: Self-reported number of days of heavy episodic drinking (4+ drinks for females/5+ drinks for males) in the past two weeks
Time Frame: Baseline, 1-month follow-up, 6-month follow-up, and 12-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Assessment-only Control | Mobile Alcohol Expectancy Intervention
Number analyzed (Participants) | 203 | 205
Number of days
  Baseline | 2.85 (2.22) | 2.85 (2.13)
  1-month follow-up: number analyzed (Participants) | 189 | 191
  1-month follow-up | 2.26 (2.32) | 1.87 (1.95)
  6-month follow-up: number analyzed (Participants) | 184 | 169
  6-month follow-up | 2.07 (2.20) | 2.04 (2.37)
  12-month follow-up: number analyzed (Participants) | 179 | 174
  12-month follow-up | 2.03 (2.13) | 1.83 (2.02)
Statistical Analysis 1: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 1-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.04, Generalized linear mixed model; Models controlled for sex, age, and college type (2-year vs. 4-year) and used a Poisson error distribution; Count/Rate Ratio = 0.83, 95% CI 2-sided [0.69 to 0.99]
Statistical Analysis 2: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 6-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.84, Generalized linear mixed model; Models controlled for sex, age, and college type (2-year vs. 4-year) and used a Poisson error distribution; Count/Rate Ratio = 0.98, 95% CI 2-sided [0.77 to 1.23]
Statistical Analysis 3: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 12-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 3]; p = 0.34, Generalized linear mixed model; Models controlled for sex, age, and college type (2-year vs. 4-year) and used a Poisson error distribution; Count/Rate Ratio = 0.90, 95% CI 2-sided [0.73 to 1.22]

4. Primary Outcome: Brief Young Adult Alcohol Consequences Questionnaire
Description: Total sum score on the Brief Young Adult Alcohol Consequences Questionnaire based on number of self-reported alcohol-related consequences experienced in the past month (range from 0-24 consequences). Higher scores indicate reporting greater number of negative alcohol-related consequences.
Time Frame: Baseline, 1-month follow-up, 6-month follow-up, and 12-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of consequences
Arm/Group | Assessment-only Control | Mobile Alcohol Expectancy Intervention
Number analyzed (Participants) | 203 | 205
number of consequences
  Baseline | 9.14 (3.82) | 8.88 (4.12)
  1-month follow-up: number analyzed (Participants) | 189 | 192
  1-month follow-up | 5.92 (4.41) | 5.85 (5.17)
  6-month follow-up: number analyzed (Participants) | 183 | 169
  6-month follow-up | 5.95 (4.93) | 5.16 (4.70)
  12-month follow-up: number analyzed (Participants) | 178 | 175
  12-month follow-up | 5.97 (4.58) | 5.89 (4.78)
Statistical Analysis 1: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 1-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.78, Generalized linear mixed model; Models controlled for sex, age, and college type (2-year vs. 4-year) and used a Poisson error distribution; Count/Rate Ratio = 0.98, 95% CI 2-sided [0.82 to 1.16]
Statistical Analysis 2: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 6-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p = 0.27, Generalized linear mixed model; Models controlled for sex, age, and college type (2-year vs. 4-year) and used a Poisson error distribution; Count/Rate Ratio = 0.90, 95% CI 2-sided [0.75 to 1.08]
Statistical Analysis 3: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 12-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — [test comment as in outcome 1, analysis 3]; p = 0.95, Generalized linear mixed model; Models controlled for sex, age, and college type (2-year vs. 4-year) and used a Poisson error distribution; Count/Rate Ratio = 1.01, 95% CI 2-sided [0.84 to 1.20]

5. Secondary Outcome: Alcohol Use Disorder Identification Test Total Score
Description: Measure of hazardous/harmful drinking in the past year based on indicators of alcohol use disorder (Total score range: 0-40, with higher values indicating greater hazardous/harmful drinking)
Time Frame: Baseline and 12-month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assessment-only Control | Mobile Alcohol Expectancy Intervention
Number analyzed (Participants) | 203 | 205
units on a scale
  Baseline: number analyzed (Participants) | 203 | 203
  Baseline | 12.52 (5.46) | 11.88 (4.87)
  12-month follow-up: number analyzed (Participants) | 177 | 171
  12-month follow-up | 10.72 (5.68) | 10.04 (5.34)
Statistical Analysis 1: Comparison: Assessment-only Control vs Mobile Alcohol Expectancy Intervention; Changes from Baseline to 12-Month Follow-Up for intervention versus assessment-only control reported in this section; Test type: Superiority — Generalized linear model was estimated using a sample of N=346; p = 0.69, Generalized linear mixed model; Model controlled for sex, age, and college type (2-year vs. 4-year) and used a negative binomial error distribution; Count/Rate Ratio = 0.98, 95% CI 2-sided [0.89 to 1.08]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between initial screening and final follow-up for each participant, a period of up to fifteen months.
Description: We used clinicaltrials.gov definitions for adverse events and serious adverse events.
Arm/Group | Assessment-only Control | Mobile Alcohol Expectancy Intervention
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/205
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/205
Other Adverse Events (participants affected / at risk) | 0/203 | 0/205

LIMITATIONS AND CAVEATS:
Nearly all study data (including all outcome data) were collected during the COVID-19 pandemic, which may have impacted alcohol expectancies and alcohol use, as well as contexts of alcohol use among young adult participants. All findings are based on self-report of alcohol use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT04213846/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT04213846/SAP_001.pdf